CLINICAL TRIAL: NCT06250023
Title: Early Shift to Oral Antibiotic Treatment for Pyogenic Vertebral Osteomyelitis (SAVE) - a Open Label Non-inferiority Nation-wide Study
Brief Title: SAVE- Oral Antibiotics for Treatment of Vertebral Osteomyelitis
Acronym: SAVE
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Anne-Mette Lebech, Consultant, associate professor, MD Dsc, Rigshospitalet, Denmark
Other Study IDs: 2023-507617-96-01
Record Dates: First submitted 2023-11-29; First posted 2024-02-08 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Osteomyelitis; Vertebra
MeSH Terms: conditions — Osteomyelitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standart of care: Standard of care (comparator)
  * Uncomplicated PVO: 2 weeks IV ABs followed by oral ABs for 4 weeks.
  * Complicated PVO: 2-4 weeks IV ABs followed by oral ABs for 8 weeks.
- Early shift: Early shift to oral ABs (intervention)
  * Uncomplicated PVO: 1 week IV ABs followed by 5 weeks of oral ABs.
  * Complicated PVO: 1 week IV ABs followed by 11 weeks of oral ABs.
  Interventions: Other: Early shift til oral antibiotic treatment for osteomyelitis

INTERVENTIONS:
Other: Early shift til oral antibiotic treatment for osteomyelitis — To investigate whether early transition to oral AB treatment after one week of IV treatment is non-inferior to the current national guideline of continued IV AB treatment for two to four weeks followed by oral AB treatment for PVO.
  Groups: Early shift

SUMMARY:
Background The current Danish National Guideline for treatment of pyogenic vertebral osteomyelitis (PVO) recommends 6 weeks antibiotic (AB) treatment, with a 2-week intravenous (IV) AB lead-in followed by 4 weeks oral AB for uncomplicated PVO, and 12 weeks AB treatment with a 2-4-week IV AB lead-in followed by 8 weeks oral AB for complicated PVO.

The primary objective of the current study is to investigate whether shortening the duration of IV AB to one week for both complicated and uncomplicated PVO is non-inferior to the current Danish National Guideline.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Diagnosed with PVO by a physician based on clinical symptoms and findings consistent with PVO in combination with diagnostic imaging (MRI, PET/CT or PET/MRI)
3. The physician responsible for the patient decides to treat the patient for PVO
4. At time of randomization CRP has decreased to < 75% of peak value or to < 20 mg/l
5. At the time of randomization patient has received maximum 7 days of appropriate IV AB for PVO -

Exclusion Criteria:

1. Previous episodes of PVO within the past 24 months
2. Spinal implants inserted prior to current episode of PVO
3. Hypersensitivity to an AB intended for use in the patient and no alternative drugs available.
4. Oral ABs not possible due to suspicion of reduced absorption
5. Oral Abs not possible due to verified or expected bacterial susceptibility or due to expected toxicity of available regimen
6. Identification of fungus, mold, TB, Brucella, Actinomyces, Nocardia and P. aeruginosa as etiology
7. Severe immunocompromise defined as primary immunodeficiencies, uncontrolled HIV/AIDS, organ transplant recipients, hematological malignancies, patients undergoing biological therapy or chemotherapy and patients treated with prednisolone >=20 mg daily >14 days
8. Verified or expected reduced compliance (for example iv drug use)
9. Pregnancy
10. Breastfeeding
11. Women of childbearing potential, who at the time of inclusion are not using and/or who will not use an effective anticonception method during the treatment period.
12. Patients not capable of providing informed consent at time of screening for inclusion
13. Diagnosed or suspected concomitant or unrelated infections necessitating IV AB therapy beyond 7 days of duration at the time of randomization -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be a nationwide, multicenter, investigator initiated, randomized, controlled, parallel group, open label, non-inferiority trial.
  The study will be conducted at departments of infectious diseases in Denmark and in collaboration with spinal surgery units carrying out infection-related spinal surgery.
  All patients diagnosed with PVO will be assessed for eligibility. Patients will be eligible for inclusion if they fulfill all the inclusion and none of the exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 530 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | Six months after completion of oral antibiotic treatment
  All-cause mortality
Primary outcome | Six months after completion of oral antibiotic treatment
  Unplanned surgical intervention in relation to the spine
Primary outcome | Six months after completion of oral antibiotic treatment
  Relapse of bacteremia with primary pathogen
Primary outcome | Six months after completion of oral antibiotic treatment
  Relapse of bacteria with the initial pathogen being cultured from relevant material from infected areas in relation to the spine or iliopsoas muscle (detected by culture)
Primary outcome | Six months after completion of oral antibiotic treatment
  Renewed course of intravenous antibiotic given for more than 7 days for treatment of pyogenic vertebral osteomyelitis

SECONDARY OUTCOMES:
Secondary outcome 1 | Six months after completion of oral antibiotic treatment
  Occurrence of each component of the composite primary endpoint from the time of shift to oral AB treatment to six months after completion of oral AB treatment.
Secondary outcome 2 | Six months after completion of oral antibiotic treatment
  Median duration of hospital admission(s) from the time of shift to oral AB treatment to six months after completion of oral AB treatment (Admission defined as overnight stay at the department)
Secondary outcome 3 | Six months after completion of oral antibiotic treatment
  Number of readmissions from the time of shift to oral AB treatment to six months after completion of oral AB treatment
Secondary outcome 4 | Six months after completion of oral antibiotic treatment
  Proportion of patients receiving additional oral AB therapy beyond the duration defined in the protocol
Secondary outcome 5 | Six months after completion of oral antibiotic treatment
  Proportion of patients having early termination of allocated treatment strategy due to adverse events, patient preference, or any other reason
Secondary outcome 6 | Six months after completion of oral antibiotic treatment
  Proportion of patients experiencing complications associated with IV treatment (e.g., catheter infections, phlebitis, bleeding, venous thrombosis, need for replacement of catheter) from the time of initiation of IV treatment for PVO to six months after completion of oral AB treatment
Secondary outcome 7 | Six months after completion of oral antibiotic treatment
  Proportion of patients experiencing severe adverse events from ABs from the time of initiation of IV treatment for PVO to six months after completion of oral AB treatment
Secondary outcome 8 | Six months after completion of oral antibiotic treatment
  Proportion of patients experiencing adverse events from ABs from the time of initiation of IV treatment for PVO to six months after completion of oral AB treatment
Secondary outcome 9 | Six months after completion of oral antibiotic treatment
  Proportion of patients diagnosed with Clostridioides difficile associated diarrhea from the time of initiation of IV treatment for PVO to six months after completion of oral AB treatment
Secondary outcome 10 | Six months after completion of oral antibiotic treatment
  Quality of life scores (EQ-5D) at the following timepoints: Randomization, 1 week after the end of AB therapy, 1 month after the end of AB therapy, 6 months after the end of oral AB therapy, and 12 months after the end of oral AB therapy
Secondary outcome 11 | Six months after completion of oral antibiotic treatment
  Resource allocation/cost assessment determined by a combination of EQ5D, DALYs, Days of hospital admission and antibiotic prescribing costs
Secondary outcome 12 | Six months after completion of oral antibiotic treatment
  CRP, WBC, alkaline phosphatase and procalcitonin at randomization as well as CRP, WBC, alkaline phosphatase weekly during treatment and at week 4, 12 and 24 after completion of oral AB treatment.
Secondary outcome 13 | Six months after completion of oral antibiotic treatment
  Presence of microbial cell-free DNA in blood samples at the time of randomization and 6 months after the end of oral AB therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Infectious Diseases, Rigshospitalet, Copenhagen, Denmark, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No